CLINICAL TRIAL: NCT00718744
Title: Standardization of Chortoglyphus Arcuatus Allergenic Extract. Determination of Biological Activity in HEP Units
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorios Leti, S.L. (Industry)
Responsible Party: María José Gómez, Laboratorios LETI S.L.Unipersonal
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2005-001194-96
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2010-08-05 (Estimated); Status verified 2010-08

CONDITIONS: Rhinitis, Allergic, Seasonal; Conjunctivitis, Allergic
Keywords: Allergen-extract; Standardization
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Conjunctivitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): In each individual patient, 10 mg/ml histamine dihydrochloride solution and a phenolated saline solution will be applied as positive and negative control respectively.
  Interventions: Other: Standardization of allergenic extract (Ch. arcuatus)

INTERVENTIONS:
Other: Standardization of allergenic extract (Ch. arcuatus) — Allergenic extract for cutaneous prick-test

SUMMARY:
The main purpose of the trial is to prove the therapeutic value of the product and enable an effective and safe dosage schedule to be recommended

DETAILED DESCRIPTION:
The skin testing procedure, based on the Nordic Guidelines is the reference method for the biological calibration of in-House Reference Preparations (IHRP). The method is not intended for routine testing of allergen extracts. The use of this procedure is the basis for the definition of biological activity units: "the activity of an allergen extract is 10,000 Biological Units (BU) per ml (10 HEP per ml), when the extract provokes an specific skin reaction in the median sensitive patient with a wheal of the same size as a wheal provoked by a positive reference solution consisting of histamine 54.3 mmol/l (for example histamine dihydrochloride 10 mg/ml), when both solutions are administrated using the same technique (prick testing) on at least 20 individuals who are clinically allergic and cutaneously reactive to the allergen concerned".

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed informed consent form by the patient
* Patients should live in a geographic zone where allergy caused by Chortoglyphus arcuatus is a relevant problem.
* Patients should not be excluded due to low or high sensitivity to the allergen, when they otherwise fulfil the inclusion criteria.
* A positive case history with inhalant allergy related to exposure to the allergen to be tested.
* A positive prick test (mean wheal diameter > 3 mm) when tested with a standardized extract prepared from the allergen source in question and/or a positive test for specific IgE.
* A mean wheal diameter > 7 mm2 obtained in a prick test with histamine dihydrochloride 10 mg/ml.
* Age: 18-50 years.
* Both genders

Exclusion Criteria:

* Immunotherapy in the past 2 years with an allergen preparation known to interfere with the allergens to be tested.
* Use of drugs that may interfere with the skin reactions.
* Pregnancy
* Dermographism
* Atopic dermatitis (locally at the test site)
* Urticaria.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-06; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Wheal size area (mm2) of the immediate phase reaction. | 30 minutes per subject

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Boquete, MD, Principal Investigator
Locations (1):
- Hospital "Xeral de Calde", Calde, Lugo, Spain